CLINICAL TRIAL: NCT01237327
Title: Follow-up of the Study 971-ONC-0028-080: Exemestane Versus Megestrol Acetate In Postmenopausal Patients With Metastatic Breast Cancer, Failing Anti-Estrogens: An Open-Label, Randomized, Parallel-Group, Phase III Comparative Study
Brief Title: Multicenter Follow Up Study Of Subjects Who Participated In An Original Protocol Of Exemestane Vs. Megestrol Acetate In Postmenopausal Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 971-ONC-0028-094; A5991027
Record Dates: First submitted 2010-11-03; First posted 2010-11-09 (Estimated); Results first posted 2011-03-14 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Advanced; Postmenopausal; Exemestane vs Megestrol
MeSH Terms: conditions — Breast Neoplasms | interventions — Megestrol Acetate; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Megestrol acetate
- 2 (Experimental)
  Interventions: Drug: exemestane (Aromasin)

INTERVENTIONS:
Drug: Megestrol acetate — Megestrol Acetate 160 mg oral tablets Qd
  Other Names: Megace
  Arms: 1
Drug: exemestane (Aromasin) — exemestane (Aromasin) 25 mg oral tablets Qd
  Other Names: Aromasin
  Arms: 2

SUMMARY:
Long term efficacy of exemestane as compared to megestrol acetate in the treatment of women with natural or induced postmenopausal status with advanced breast cancer whose disease has progressed following anti-estrogens or anti-estrogens plus chemotherapy and who had participated on an original study of exemestane vs megestrol : study 971-ONC-0028-080.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in study 971-ONC-0028-080.

Exclusion Criteria:

* Subjects who had not previously participated in study 971-ONC-0028-080.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2001-11; Primary Completion 2007-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- China (7):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - PLA 307 Hospital, Beijing
  - Ba Yi Hospital, Cancer Center of CPLA, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Cancer Hospital, Shanghai
  - The 2nd Central Hospital of Tianjin, Tianjin
  - The 1st Affiliated Hospital, Xi'an Jiao Tong University, Xi'an

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=971-ONC-0028-094&StudyName=Open%20Label%20Randomized%20Controlled%20Multicenter%20Follow%20Up%20Study%20Of%20Subjects%20Who%20Participated%20In%20An%20Original%20Protocol%20Of%20Exemestane%20Vs

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Follow-up study for participants in core study who completed 26 weeks of treatment, progressed while on therapy, or dropped out for any reason. Those who benefitted from core study treatment continued according to original randomization. Those who dropped out of core study received therapy appropriate for disease and were followed for survival.
Groups:
- Exemestane: Exemestane 25 milligram (mg) oral tablet taken once daily
- Megestrol Acetate: Megestrol acetate 160 mg tablet taken once daily
Period: Overall Study
Arm/Group | Exemestane | Megestrol Acetate
Started | 43 | 41
Stopped Treatment in Core Study (D/C) | 22 (Continued in Extension Study for follow-up only; not treated with study medication.) | 24 (Continued in Extension Study for follow-up only; not treated with study medication.)
Completed Treatment in Core Study | 3 (Completed 26 weeks of treatment in Core Study; continued in Extension Study for follow-up only.) | 2 (Completed 26 weeks of treatment in Core Study; continued in Extension Study for follow-up only.)
Continued Treatment in Extension Study | 21 | 17
Completed | 1 (On treatment at Extension Study cut-off date.) | 1 (On treatment at Extension Study cut-off date.)
Not Completed | 42 | 40
Not completed — Protocol Violation: Core Study | 1 | 0
Not completed — Completed 26 weeks treatment:Core Study | 3 | 2
Not completed — Progression of Disease: Core Study | 18 | 22
Not completed — Progression of Disease: Extension Study | 15 | 13
Not completed — Protocol Specific Withdrawal Criteria | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane | Megestrol Acetate | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Customized [Number; unit: participants]
  < 50 years | 10 | 15 | 25
  50 to 64 years | 17 | 24 | 41
  65 to 79 years | 16 | 2 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 84
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival in months measured from date of starting treatment in core study to date of death for any reason.
Time Frame: Every 12 weeks up to 6 years
Population: Intent-to-treat (ITT): participants randomized to study medication in core study who consented to participation in extension study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane | Megestrol Acetate
Number analyzed (Participants) | 43 | 41
months | 29.2 [22.9 to 47.8] | 16.3 [11.6 to 27.6]
Statistical Analysis 1: Comparison: Exemestane vs Megestrol Acetate; Overall survival compared using the hazard ratio; hazard ratio <1.0 is in favor of exemestane; Test type: Superiority or Other; p = 0.3348, Log Rank; Hazard Ratio (HR) = 0.7799, 95% CI 2-sided [0.47 to 1.294]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Percentage of participants achieving an objective response (OR) defined as complete response (CR) or partial response (PR) out of the total number of participants randomized in each treatment group
Time Frame: Every 12 weeks up to 6 years
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Exemestane | Megestrol Acetate
Number analyzed (Participants) | 43 | 41
percentage of participants | 23.3 | 12.2

3. Secondary Outcome: Duration of Response (DR)
Description: Duration of objective response (complete response [CR] or partial response [PR]) calculated from date objective response was first documented to date of progressive disease. For subjects proceeding from PR to CR, the onset of PR was taken as the onset of objective response.
Time Frame: Every 12 weeks up to 6 years
Population: ITT.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane | Megestrol Acetate
Number analyzed (Participants) | 43 | 41
months | 12.9 [10.8 to 49.0] | 35.4 [23.6 to NA] — The upper limit of the 95% confidence interval for the megestrol acetate treatment group was inestimable and is shown as N/A.because not enough participants progressed from objective response to progressive disease during the study period.

4. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP = time between first day of study treatment and date of documented disease progression, or date of tumor-related death in the absence of previously documented progressive disease (PD). PD defined as a 25% or greater increase in size of 1 or more lesions compared to smallest previous assessment, or appearance of new lesion, or unequivocal worsening of bone lesions, or progression of nonevaluable lesions.
Time Frame: Every 12 weeks up to 6 years
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane | Megestrol Acetate
Number analyzed (Participants) | 43 | 41
months | 6.0 [3.7 to 13.0] | 3.7 [2.1 to 8.9]

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF = time between first day of study treatment and date of diagnosis of progression, withdrawal from study treatment for any reason, administration of other antitumor treatment, or death from any cause, whichever was the earliest event.
Time Frame: Every 12 weeks up to 6 years
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane | Megestrol Acetate
Number analyzed (Participants) | 43 | 41
months | 6.0 [3.7 to 11.4] | 3.7 [2.1 to 8.8]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Exemestane | Megestrol Acetate
Serious Adverse Events (participants affected / at risk) | 1/41 | 2/40
Other Adverse Events (participants affected / at risk) | 24/41 | 25/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=41) | Megestrol Acetate (N=40)
Chest pain NEC (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Headache NOS (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=41) | Megestrol Acetate (N=40)
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 2
Chest pain NEC (General disorders) | 1 | 2
Fatigue (General disorders) | 1 | 6
Pain NOS (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Influenza (Infections and infestations) | 3 | 1
Aspartate aminotransferase (Investigations) | 1 | 1
Weight increased (Investigations) | 3 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Face eodema (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Sweating increased (Skin and subcutaneous tissue disorders) | 5 | 4
Flushing (Vascular disorders) | 5 | 0
Oedema NOS (Cardiac disorders) | 0 | 2
Tachycardia NOS (Cardiac disorders) | 0 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chest mass NOS (General disorders) | 0 | 1
Oedema NOS (General disorders) | 0 | 1
Infection NOS (Infections and infestations) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase (Investigations) | 0 | 1
Gamma-glutamyltransferase (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Diabetes mellitus NOS (Metabolism and nutrition disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (exc vertigo) (Nervous system disorders) | 0 | 2
Headache NOS (Nervous system disorders) | 0 | 1
Insomnia NEC (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Mood alteration NOS (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1
Breast mass NOS (Reproductive system and breast disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
At the time of study completion in 2007, via protocol amendment participants still on treatment were allowed to continue treatment, being monitored for Serious Adverse Events (SAE) only. The final participant discontinued in 2009.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.